CLINICAL TRIAL: NCT00047060
Title: A Phase I/II Study of HLA-matched Mobilized Peripheral Blood Hematopoietic Stem Cell Transplantation for Advanced Mycosis Fungoides/Sezary Syndrome Using Nonmyeloablative Conditioning With Campath-1H
Brief Title: Stem Cell Transplant Therapy With Campath-1H for Treating Advanced Mycosis Fungoides and Sezary Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020250; 02-H-0250 (Other: NIH - National Heart, Lung, and Blood Institute); NCT00042640 (obsolete NCT alias)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2019-02-13

CONDITIONS: Mycosis Fungoides; Sezary Syndrome
Keywords: Cutaneous T Cell Lymphoma; Allogeneic PBSCT; Low Intensity Regimen; Mycosis Fungoides; Sezary Syndrome; CTCL
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — Cyclosporine; fludarabine; fludarabine phosphate; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Stem Cell Transplant Therapy With Campath-1H (Experimental): Recipients received a nonmyeloablative preparative regimen of alemtuzumab 30mg iv three times a week for two weeks followed by fludarabine 25mg/m2/day for five days followed by a PBPC graft targeted to deliver ≥ 5x106 CD34+ cells/kg. Cyclosporine A (CSA) for GVHD prophylaxis used initially with target CSA levels in the therapeutic range (200 -400 ng/ml).
  Interventions: Other: A matched peripheral donor stem cells; Drug: cyclosporine; Drug: fludarabine; Drug: Campath

INTERVENTIONS:
Other: A matched peripheral donor stem cells — A matched peripheral donor stem cells
  Other Names: Allogeneic peripheral stem cell transplant
Drug: cyclosporine — cyclosporine
  Other Names: CSA
Drug: fludarabine — fludarabine
  Other Names: fludara
Drug: Campath — Campath
  Other Names: Alemtuzumab

SUMMARY:
This study will investigate the safety and effectiveness of a modified donor stem cell transplantation procedure for treating advanced mycosis fungoides (MF), a lymphoma primarily affecting the skin, and Sezary syndrome (SS), a leukemic form of the disease. Donated stem cells (cells produced by the bone marrow that mature into the different blood components white cells, red cells and platelets) can cure patients with certain leukemias and lymphomas and multiple myeloma. These cells generate a completely new, functioning bone marrow. In addition, immune cells from the donor grow and generate a new immune system to help fight infections. The new immune cells also attack any residual tumor cells left in the body after intensive chemotherapy. However, stem cell transplantation carries a significant risk of death, because it requires completely suppressing the immune system with high-dose chemotherapy and radiation. In addition, lymphocytes from the donor may cause what is called graft vs. host disease (GvHD), in which these cells see the patient s cells as foreign and mount an immune response to destroy them. To try to reduce these risks, patients in this study will be given low-dose chemotherapy and no radiation, a regimen that is easier for the body to tolerate and involves a shorter period of complete immune suppression. In addition, a monoclonal antibody called Campath-1H will be given to target lymphocytes, including those that have become cancerous.

Patients with advanced MF or SS who are between 18 and 70 years of age and have a matched family donor 18 years of age or older may be eligible for this study. Candidates will have a medical history, physical examination and blood tests, lung and heart function tests, X-rays of the chest, eye examination, and bone marrow sampling (withdrawal through a needle of about a tablespoon of marrow from the hip bone), and small skin biopsy (surgical removal of a piece of tissue for microscopic examination) or needle biopsy of the tumor.

Stem cells will be collected from both the patient and donor. To do this, the hormone G-CSF will be injected under the skin for several days to push stem cells out of the bone marrow into the bloodstream. Then, the stem cells will be collected by apheresis. In this procedure the blood is drawn through a needle placed in one arm and pumped into a machine where the required cells are separated out and removed. The rest of the blood is returned through a needle in the other arm.

Before the transplant, a central venous line (large plastic tube) is placed into a major vein. This tube can stay in the body and be used the entire treatment period to deliver the donated stem cells, give medications, transfuse blood, if needed, and withdraw blood samples. Several days before the transplant procedure, patients will start a conditioning regimen of low-dose chemotherapy with Campath 1H, fludarabine, and, if necessary, cyclophosphamide. When the conditioning therapy is completed, the stem cells will be infused over a period of up to 4 hours. To help prevent rejection of donor cells and GvHD, cyclosporine and mycophenolate mofetil will be given by mouth or by vein for about 3 months starting 4 days before the transplantation.

The anticipated hospital stay is 3 to 4 days, when the first 3 doses of Campath will be monitored for drug side effects. The rest of the procedures, including the transplant, can be done on an outpatient basis. Follow-up visits for the first 3 months after the transplant will be scheduled once or twice a week for a physical examination, blood tests and symptoms check. Then, visits will be scheduled at 6, 12, 18, 24, 30, 36, and 48 months post-transplant. Visits for the first 3 years will include blood tests, skin biopsies, and bone marrow biopsies.

DETAILED DESCRIPTION:
Primary cutaneous T-cell lymphomas (CTCL) are a group of lymphoproliferative disorders characterized by localization of neoplastic T cells to the skin at presentation. Mycosis fungoides (MF) and its leukemic variant Sezary syndrome (SS) are the most prevalent forms of CTCL. While early stage MF is restricted to patches and plaques involving the skin, most patients eventually develop cutaneous tumors, generalized erythroderma, or dissemination to peripheral blood, lymph nodes or visceral organs. Currently existing therapy of tumor-stage and disseminated CTCL is palliative, with most patients dying within 1-5 years. The presence of CD8+ cells in close proximity to dermal neoplastic infiltrates in early stages of the disease, and the clinical response seen with some immunomodulatory agents suggests that CTCL may be potential targets for immunotherapy-based interventions.

Allogeneic stem cell transplantation is a curative treatment modality successfully employed in a number of hematologic malignancies. The curative effect of this approach is in part mediated by donor-derived T lymphocytes with reactivity for patient leukemic cells. The power of this graft versus leukemia effect (GVL) is best illustrated in patients with relapsed Chronic Myeloid Leukemia (CML) after an allogeneic bone marrow transplant, in whom a single donor lymphocyte infusion (DLI) can induce remission. We hypothesize that neoplastic T cells in MF/SS may similarly be susceptible to a graft vs. tumor (GVT) effect. Unfortunately, advanced patient age and a 25% to 35% risk of transplant related mortality (TRM) preclude the use of conventional 'dose- intensive' allogeneic peripheral blood stem cell transplantation (PBSCT) in patients with advanced CTCL who might otherwise benefit from this approach. The risk of TRM related to conditioning can be circumvented at least partially by using a reduced-intensity conditioning regimen to prepare the patient for transplantation.

In this study, we will treat male and non-pregnant female subjects between the ages of 18 and 70 years (both inclusive) suffering from advanced MF/SS with an allogeneic peripheral blood stem cell (PBSC) transplant from an HLA-matched family donor or an HLA matched (10/10 allele level match) unrelated donor. A low intensity, nonmyeloablative conditioning regimen employing the anti-CD52 monoclonal antibody Campath-1H (alemtuzumab) and fludarabine will be used to induce host immunosuppression to facilitate donor hematopoietic and lymphoid engraftment. We anticipate minimal host myelosuppression and consequently reduced early transplant toxicity with this conditioning regimen. Immune and hematopoietic reconstitution will be achieved by infusion of unmanipulated donor-derived granulocyte colony stimulation factor (G-CSF) mobilized peripheral blood stem cells. Infusion of donor lymphocytes in incremental doses will be used to promote engraftment or disease regression when indicated. Cyclosporine A (CSA) will be used as prophylaxis against graft vs host disease (GVHD), with dose adjustments made as necessary to favor complete donor chimerism and disease regression.

A total of up to 25 subjects (transplant recipients) will be treated on this protocol. The primary end point of this study is efficacy (proportion of subjects achieving a complete response). Other end points include assessment of donor-host chimerism in various hematopoietic and lymphoid cells, overall response, incidence of acute and chronic GVHD, graft failure, assessment of lymphoid subset reconstitution, transplant related morbidity and mortality and disease-free and overall survival and the outcomes of transplantation by the donor type (related vs. unrelated).

ELIGIBILITY:
* INCLUSION CRITERIA-RECIPIENT:

Ages 18-70 years (both inclusive)

Stages IIb to IVb patients with MF (biopsy diagnostic or consistent with MF) who have progressed despite at least one treatment regimen and all patients with SS

AND

Anticipated median survival less than 5 years or debilitation as a result of their disease.

Recovery from acute toxicity of prior treatment for MF/SS (to less than or equal to grade 1 [CTCAE v3.0]) or stabilization of toxicity occurring from prior therapy for MF/SS.

HIV negative

ECOG performance status of 1 or less.

No major organ dysfunction precluding transplantation.

DLCO greater than or equal to 60 percent predicted

Left ventricular ejection fraction greater than or equal to 40 percent.

Less than or equal to 25 percent of liver involved with metastatic tumor by CT scan.

6/6 HLA matched family donor or 10/10 matched unrelated donor at the allelic level available

Ability to comprehend the investigational nature of the study and provide informed consent.

INCLUSION CRITERIA-RELATED and UNRELATED DONOR:<TAB>

6/6 HLA- matched family donor or 10/10 HLA-matched unrelated donor

Age greater than or equal to 18 years

Ability to comprehend the investigational nature of the study and provide informed consent.

For unrelated donor, the NMDP unrelated donor inclusion criteria will be used as outlined in document (http://bethematch.org/WorkArea/DownloadAsset.aspx?id=1960).

Donor eligibility will be completed per NMDP standards and in accordance with most recent and stringent FDA guidelines.

EXCLUSION CRITERIA (ANY OF THE FOLLOWING)-RECIPIENT

Patient pregnant or lactating

Age greater than 70 or less than 18 years

ECOG performance status of 2 or more.

Psychiatric disorder or mental deficiency of the recipient or donor sufficiently severe as to make compliance with the BMT treatment unlikely and making informed consent impossible.

Major anticipated illness or organ failure incompatible with survival from BMT and where survival is considered insufficient to assess transplant outcome (i.e. less than 3 months).

DLCO less than 60 percent predicted

Left ventricular ejection fraction less than 40 percent

Serum creatinine greater than 2.0 mg/dl

Serum bilirubin greater than 4 mg/dl, transaminases greater than 5 times the upper limit of normal

HIV positive

History of other malignancies in the last five years with the exception of basal cell or squamous cell carcinoma of the skin

Evidence for CNS metastatic disease

Disease involving greater than 25 percent of the liver radiographically.

EXCLUSION CRITERIA (any of the following)-RELATED AND UNRELATED DONOR:

Donor pregnant or lactating

Age less than 18 years

HIV positive (donors who are positive for hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV-1) will be used at the discretion of the investigator following counseling and approval from the recipient).

Sickling hemoglobinopathy including HbSS or HbsC (for unrelated donors, testing for hemoglobinopathies will only be done when clinically indicated).

History of malignancy within 5 years except basal cell or squamous carcinoma of the skin.

Donor unfit to receive G-CSF and undergo apheresis (Uncontrolled hypertension, history of stroke, thrombocytopenia).

Psychiatric disorder or mental deficiency of the donor sufficiently severe as to make compliance with the BMT treatment unlikely and making informed consent impossible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2002-07-30; Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Aue, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Siegel RS, Pandolfino T, Guitart J, Rosen S, Kuzel TM. Primary cutaneous T-cell lymphoma: review and current concepts. J Clin Oncol. 2000 Aug;18(15):2908-25. doi: 10.1200/JCO.2000.18.15.2908. PMID 10920140
- [Background] Diamandidou E, Cohen PR, Kurzrock R. Mycosis fungoides and Sezary syndrome. Blood. 1996 Oct 1;88(7):2385-409. No abstract available. PMID 8839829
- [Background] Rook AH, Heald P. The immunopathogenesis of cutaneous T-cell lymphoma. Hematol Oncol Clin North Am. 1995 Oct;9(5):997-1010. PMID 8522492
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-H-0250.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Stem Cell Transplant Therapy With Campath-1H: Subjects received a nonmyeloablative preparative regimen of alemtuzumab 30mg IV three times a week for two weeks followed by fludarabine 25mg/m^2/day for five days followed by a PBPC graft targeted to deliver ≥ 5x10^6 CD34+ cells/kg. Cyclosporine A (CSA) for GVHD prophylaxis will be used initially with target CSA levels in the therapeutic range (200-400 ng/ml)
Period: Overall Study
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Started | 5
Completed | 3
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Nonmyeloablative Preparative Regimen
Description: Proportion of subjects achieving a complete response. Complete response (CR) is defined as: disappearance of all signs and symptoms of cutaneous T-cell lymphomas (CTCL) for a period of at least one month.
Time Frame: 36 months
Population: Received a nonmyeloablative preparative regimen of alemtuzumab 30mg IV 3x a week for 2 weeks followed by fludarabine 25mg/m^2/day for five days followed by a PBPC graft targeted to deliver ≥ 5x10^6 CD34+ cells/kg. Cyclosporine A (CSA) for GVHD prophylaxis will be used initially w/target CSA levels in the therapeutic range (200 -400 ng/ml).
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants | 4

2. Secondary Outcome: Number of Participants Who Experienced Acute GVHD Grades II-IV
Description: Number of participants who experienced acute GVHD grades II-IV
  Acute-GVHD was graded and staged prospectively using criteria from the 1994 Consensus Conference on Acute- GVHD Grading.
  Grades are defined as:
  Grade II: Skin = rash on 25-50 percent body surface area; Liver = Total Bilirubin 3.1-6.0 mg/dL; Lower GI = Diarrhea 1001-1500 mL/day.
  Grade III: Skin = Rash on >50% of body surface; Liver = Total Bilirubin 6.1 - 15.0 mg/dL; Lower GI = Diarrhea > 1500 mL/day.
  Grade IV: Skin = Generalized erythroderma plus bullous formation; Liver = Total Bilirubin >15 mg/dL; Lower GI = Severe abdominal pain with or without ileus.
  Grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: up to 100 days
Measure: Count of Participants; unit: Participants
Groups:
- Stem Cell Transplant Therapy With Campath-1H: Subjects received a nonmyeloablative preparative regimen of alemtuzumab 30mg iv three times a week for two weeks followed by fludarabine 25mg/m^2/day for five days followed by a PBPC graft targeted to deliver ≥ 5x10^6 CD34+ cells/kg. Cyclosporine A (CSA) for GVHD prophylaxis will be used initially with target CSA levels in the therapeutic range (200 -400 ng/ml).
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants
  Grade II | 0
  Grade III-IV | 1

3. Secondary Outcome: Number of Participant Who Experienced Chronic Graft Versus Host Disease
Description: Number of participant who experienced chronic graft versus host disease (GVHD) following stem cell transplant The diagnosis of clinical features of chronic-GVHD was determined prospectively and classified retrospectively into limited or extensive based on the Revised Seattle Classification. Chronic GvHD severity categorized as "limited" is defined as: localized skin lesions with or without limited hepatic involvement and "extensive" is defined as: generalized skin involvement, major hepatic complications, or involvement of any other organ.
Time Frame: Day 100 up to 3 years
Population: The analyses included only those participants that engrafted and survived over 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants
  Limited | 3
  Extensive | 0

4. Secondary Outcome: Number of Participants That Experienced Graft Failure
Description: Number of participants that experienced graft failure. Graft failure is defined as: the failure to achieve sustained engraftment following stem cell transplantation.
Time Frame: up to 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants | 0

5. Secondary Outcome: Overall Response
Description: Overall response following stem cell transplant. Complete response (CR) is defined as: disappearance of all signs and symptoms of cutaneous T-cell lymphomas (CTCL) for a period of at least one month.
  Partial response (PR) - a 50% or greater decrease in the sum of the products of the longest perpendicular diameters of all measured lesions (a greater than 50% reduction in area of disease involvement in the case of cutaneous disease) lasting for a period of at least one month. No new metastatic lesions may appear.
  Stable disease is defined as: tumor measurements not meeting the criteria of CR, PR, or PD.
  Progressive disease (PD) - increase of 25% or greater in the sum of the products of the longest perpendicular diameters of all measured lesions (a greater than 25% increase in area of disease involvement in the case of cutaneous disease) compared to the smallest previous measurements, or the development of any new metastatic or cutaneous disease.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants
  Complete Response (CR) | 4
  Stable Disease | 1
  Partial response (PR) | 0
  Progressive disease (PD) | 0

6. Secondary Outcome: Number of Participants Who Experienced Transplant Related Mortality
Description: Number of Participants who experienced transplant related mortality by day 100
Time Frame: day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants | 0

7. Secondary Outcome: Number of Participants Overall Survival
Description: Number of participants overall survival following stem cell transplant. Overall survival is defined as number participants alive following stem cell transplant
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants | 3

8. Secondary Outcome: Number of Participants That Remained Disease-free
Description: Number of participants that remained Disease-free survival following stem cell transplant. Disease-free survival is defined as survival free of disease relapse or disease progression following stem cell transplant.
Time Frame: up to 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants | 4

9. Secondary Outcome: Number of Participants That Experienced Engraftment
Description: Number of participants that experienced engraftment following stem cell transplant. Engraftment is defined as neutrophil count is greater than 0.5 x10^9.
Time Frame: up to 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants | 5

10. Secondary Outcome: Number of Participants That Experienced Platelet Recovery
Description: Number of participants that experienced platelet recovery up to day 100 following stem cell transplant. Platelet recovery is defined as platelet count is greater than 50 x 10^9/l without platelet transfusion.
Time Frame: up to 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants | 5

11. Secondary Outcome: Number of Participants That Experienced Red Blood Cell Recovery
Description: Number of participants that experienced red blood cell recovery following stem cell transplant. Red blood cell recovery is defined as achieving transfusion independence.
Time Frame: up to 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
Participants | 5

12. Secondary Outcome: Median Time in Months to Achieve Full Myeloid and Full Donor T-cell Chimerism
Description: Median time in months to achieve full myeloid and full donor T-cell Chimerism. Myeloid (CD34+) and T-cell (CD3+) chimerisms were determined by PCR analysis of short tandem repeats (STR). Full donor chimerism is defined as >95% donor- derived cells in the peripheral blood in a specific lineage.
Time Frame: Up to 22 months
Measure: Median (Full Range); unit: months
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
Number analyzed (Participants) | 5
months
  Myeloid Chimerism | 9 [3 to 18]
  Donor T-cell Chimerism | 7 [4 to 22]

ADVERSE EVENTS:
Time Frame: Up to 13 years
Groups:
- Stem Cell Transplant Therapy With Campath-1H: Subjects received a nonmyeloablative preparative regimen of alemtuzumab 30mg iv three times a week for two weeks followed by fludarabine 25mg/m2/day for five days followed by a PBPC graft targeted to deliver ≥ 5x106 CD34+ cells/kg. Cyclosporine A (CSA) for GVHD prophylaxis will be used initially with target CSA levels in the therapeutic range (200 -400 ng/ml).
Arm/Group | Stem Cell Transplant Therapy With Campath-1H
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 5/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stem Cell Transplant Therapy With Campath-1H (N=5)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Eyelid disorder (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disease Progression (General disorders) | 2
Fatigue (General disorders) | 1
Pain (General disorders) | 2
Acute graft versus host disease (Immune system disorders) | 1
chronic graft versus host disease (Immune system disorders) | 1
Candida infection (Infections and infestations) | 1
Cytomegalovirus syndrome (Infections and infestations) | 3
Herpes Zoster (Infections and infestations) | 1
influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Haematological malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Headache (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT00047060/Prot_SAP_000.pdf